CLINICAL TRIAL: NCT00252603
Title: Galantamine Versus Placebo in Childhood Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Alliance for Autism Research (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4682
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Autism; Childhood Autism
Keywords: Autism; Childhood Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
Autism is a severe neurodevelopmental disorder that affects up to 16 in 10,000 individuals. It is a pervasive developmental disorder affecting social, communicative, and compulsive/repetitive behaviors characterized by stereotypic complex hand and body movements, craving for sameness, and narrow repetitive interests. Autism severely impacts both the affected individual and family members.

The proposed study is designed to assess the efficacy of treatment with Galantamine vs. placebo in childhood/adolescent autism fulfilling DSM-IV and Autism Diagnostic Interview (ADI) criteria. We therefore hypothesize:

1. Galantamine will be superior to placebo in the acute treatment of global autism.
2. Galantamine will be superior to placebo in improving functional ability.
3. Galantamine will be superior to placebo in improving language function.
4. Galantamine will be superior to placebo improving irritable and hyperactive behavior.
5. Galantamine will be superior to placebo in improving social deficits.

DETAILED DESCRIPTION:
Once enrolled in the study, subjects will receive evaluations and testing to determine if they meet the necessary criteria for admission into study treatment. Subjects will not be responsible for the costs of any evaluations or tests conducted as part of this study.

First, subjects will receive a psychiatric and medical evaluation by the study psychiatrist to see if she/he has any psychiatric or medical illnesses that would interfere with their ability to participate in this study. These evaluations may take up to an hour to complete. In addition, subjects will be asked to participate in a psychiatric interview designed to determine the child's diagnosis and current problem areas. The subject's parent will also be asked to fill out psychiatric questionnaires. The interview and questionnaires may take up to 4 hours to complete.

Second, urine and blood samples will be needed for routine tests two times during this study (before any study related tests are done, and at the end of the study). Two teaspoons of blood will be drawn each time. The urine sample will be analyzed in order to assess kidney function and to screen for the presence of drugs (such as cocaine, marijuana, heroin, etc.). A positive drug screen would result in the inability of the child to participate in this study. Drug screen results will be kept confidential. In addition, an electrocardiogram will be performed to determine heartbeat.

Lastly, a pregnancy test will be conducted on the urine sample if the child is female and has reached puberty. The child should not be in this study if she is pregnant or a nursing mother. A positive urine pregnancy test would cause the child to be removed from the study. If the child is sexually active, she must be using an effective method of birth control during her participation in this study. Acceptable methods of birth control are oral contraceptive medications (the administration of which must be parentally supervised), IUD, depot medication and tubal ligation.

Subjects will be assigned by chance to receive either the active medication (Galantamine) or placebo (sugar pill) for 12 weeks, much like the flip of a coin. Neither the parent/child nor the investigator will know which of the two treatments the child is receiving. The child has a 50% chance of being assigned to receive placebo during the study or the active medication, Galantamine, during the study.

The child will need to be seen weekly by the study psychiatrist for the first 4 weeks of the twelve-week study, and every other week for the remaining weeks of the study. During these visits the study psychiatrist will ask the parent for feedback on his/her child's condition and any changes that may be related to the medication, including possible side effects, such as nausea and headaches, and will check the child's condition. The psychiatrist will also record his/her weight. These study visits will generally last approximately 30 minutes.

ELIGIBILITY:
1. Meets DSM-IV, ADI-R and ADOS-G criteria for autistic disorder
2. Age 5-17 years
3. Outpatients
4. Parent or legal guardian willing to sign informed consent.
5. Male or female patients
6. Patient scores at least a "4" (moderately ill) on the Clinical Global Impression Scale for Autistic Disorder (CGI AD).
7. Children who are minimally or non- verbal as indicated by a score of 50% of an 18 month old on the MacArthur Communicative Development Inventory

Exclusion Criteria:

1. Subjects with any of the following past or present mental disorders: psychotic disorders, mood disorders, including bipolar disorders.
2. Subjects who have displayed significant self-injurious behavior (children who have caused visible harm to themselves).
3. Subjects with active seizure disorder (seizures within the past six months).
4. Subjects with clinically significant or unstable medical illness, including patients with current evidence of clinically significant hematopoietic, or cardiovascular disease.
5. Subjects with present or history of the following:

   * gastrointestinal, liver, kidney, or other known conditions which will presently interfere with the absorption, distribution, metabolism, or excretion of drugs,
   * seizure disorders (active), cerebrovascular disease or brain trauma as etiology of autistic behavior,
   * clinically significant unstable endocrine disorder, such as hypo- or hyperthyroidism or diabetes,
   * recent history or presence of any form of malignancy.
6. Subjects who report significant improvement of autism symptoms and behaviors to current medications or have only global autism ratings on the CGI of absent, minimal or mild severity, or who are more than minimally verbal.
7. Subjects whose global autism ratings are assessed as being absent, minimal or mild.
8. Treatment within the previous 30 days with any drug known to have a well-defined potential for toxicity to a major organ.
9. Subjects with clinically significant abnormalities in laboratory tests or physical exam.
10. Subjects likely to require any other psychotropic medication during the study, with the exception of clonidine for insomnia (started at least one month prior to entrance into the study), as well as anticonvulsants at a constant dose for stable seizure disorder or, unless otherwise permitted.
11. Subjects unable to tolerate taper from psychoactive medication, if specified.
12. Subjects with a history of hypersensitivity or severe side effects associated with the use of galantamine, or other acetylcholinesterase inhibitors.
13. Subjects with a history of prior treatment with galantamine of 4mg/day for 6 weeks.
14. Subjects who have received any of the following interventions within the prescribed period before starting treatment:

    * investigational drugs within the previous 30 days.
    * monoamine oxidase inhibitors within the previous fourteen days.
    * long-acting phenothiazines within the previous six weeks.
    * other psychotropic drugs within the previous seven days, unless otherwise permitted.
15. Subjects with any organic or systemic disease or patients who require a therapeutic intervention, not otherwise specified, which would confound the evaluation of the safety of the study medication.
16. Subjects who reside in a remote geographical area or who do not have regular access to transportation to the clinical facility.

Gender

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2004-04; Study Completion 2007-04

PRIMARY OUTCOMES:
Autism Diagnostic Observation Schedule-Generic (ADOS-G)- Change from Baseline to Final Visit
Clinical Global Impression Improvement (CGI)- Change from Baseline to Final Visit
Aberrant Behavior Checklist (ABC) (hyperactivity/irritability sections)- Change from Baseline to Final Visit
Vineland Adaptive Behavior Scale- Change from Baseline to Final Visit
MacArthur Communicative Development Inventory (MCDI)- Change from Baseline to Final Visit
Conners' Parent Rating Scale-Revised: Long form (CPRS-R:L)- Change from Baseline to Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Sherie Novotny, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Robert Wood Johnson Medical School - Dept of Psychiatry, Piscataway, New Jersey, United States

REFERENCES:
- [Background] Allin M, Matsumoto H, Santhouse AM, Nosarti C, AlAsady MH, Stewart AL, Rifkin L, Murray RM. Cognitive and motor function and the size of the cerebellum in adolescents born very pre-term. Brain. 2001 Jan;124(Pt 1):60-6. doi: 10.1093/brain/124.1.60. PMID 11133787
- [Background] Aman MG, Van Bourgondien ME, Wolford PL, Sarphare G. Psychotropic and anticonvulsant drugs in subjects with autism: prevalence and patterns of use. J Am Acad Child Adolesc Psychiatry. 1995 Dec;34(12):1672-81. doi: 10.1097/00004583-199512000-00018. PMID 8543539
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. Psychometric characteristics of the aberrant behavior checklist. Am J Ment Defic. 1985 Mar;89(5):492-502. PMID 3158201
- [Background] Anderson LT, Campbell M, Grega DM, Perry R, Small AM, Green WH. Haloperidol in the treatment of infantile autism: effects on learning and behavioral symptoms. Am J Psychiatry. 1984 Oct;141(10):1195-202. doi: 10.1176/ajp.141.10.1195. PMID 6385731
- [Background] Birmaher B, Quintana H, Greenhill LL. Methylphenidate treatment of hyperactive autistic children. J Am Acad Child Adolesc Psychiatry. 1988 Mar;27(2):248-51. doi: 10.1097/00004583-198803000-00020. No abstract available. PMID 3360732
- [Background] Chakrabarti S, Fombonne E. Pervasive developmental disorders in preschool children. JAMA. 2001 Jun 27;285(24):3093-9. doi: 10.1001/jama.285.24.3093. PMID 11427137
- [Background] Ghaziuddin M, Tsai L, Ghaziuddin N. Fluoxetine in autism with depression. J Am Acad Child Adolesc Psychiatry. 1991 May;30(3):508-9. doi: 10.1097/00004583-199105000-00029. No abstract available. PMID 2055895
- [Background] Greenspan, S.I. & Wieder, S. Developmental patterns and outcomes in infants and children with disorders in relating and communicating A chart review of 200 cases of children with autistic spectrum diagnoses. J Dev Learning Disord, 1997;1:87-141.
- [Background] Kern JK, Miller VS, Cauller PL, Kendall PR, Mehta PJ, Dodd M. Effectiveness of N,N-dimethylglycine in autism and pervasive developmental disorder. J Child Neurol. 2001 Mar;16(3):169-73. doi: 10.1177/088307380101600303. PMID 11305684
- [Background] Martin A, Scahill L, Klin A, Volkmar FR. Higher-functioning pervasive developmental disorders: rates and patterns of psychotropic drug use. J Am Acad Child Adolesc Psychiatry. 1999 Jul;38(7):923-31. doi: 10.1097/00004583-199907000-00024. PMID 10405512
- [Background] Perry EK, Lee ML, Martin-Ruiz CM, Court JA, Volsen SG, Merrit J, Folly E, Iversen PE, Bauman ML, Perry RH, Wenk GL. Cholinergic activity in autism: abnormalities in the cerebral cortex and basal forebrain. Am J Psychiatry. 2001 Jul;158(7):1058-66. doi: 10.1176/appi.ajp.158.7.1058. PMID 11431227
- [Background] Ritvo ER, Mason-Brothers A, Freeman BJ, Pingree C, Jenson WR, McMahon WM, Petersen PB, Jorde LB, Mo A, Ritvo A. The UCLA-University of Utah epidemiologic survey of autism: the etiologic role of rare diseases. Am J Psychiatry. 1990 Dec;147(12):1614-21. doi: 10.1176/ajp.147.12.1614. PMID 2244638
- [Background] Rutter M. The development of infantile autism. Psychol Med. 1974 May;4(2):147-63. doi: 10.1017/s0033291700041982. No abstract available. PMID 4597904
- [Background] Steffenburg S. Neuropsychiatric assessment of children with autism: a population-based study. Dev Med Child Neurol. 1991 Jun;33(6):495-511. doi: 10.1111/j.1469-8749.1991.tb14915.x. PMID 1864476
- [Background] Thal DJ, O'Hanlon L, Clemmons M, Fralin L. Validity of a parent report measure of vocabulary and syntax for preschool children with language impairment. J Speech Lang Hear Res. 1999 Apr;42(2):482-96. doi: 10.1044/jslhr.4202.482. PMID 10229462
- [Background] Voelker SL, Shore DL, Brown-More C, Hill LC, Miller LT, Perry J. Validity of self-report of adaptive behavior skills by adults with mental retardation. Ment Retard. 1990 Oct;28(5):305-9. PMID 2255260
- [Background] Woodruff-Pak DS, Vogel RW 3rd, Wenk GL. Galantamine: effect on nicotinic receptor binding, acetylcholinesterase inhibition, and learning. Proc Natl Acad Sci U S A. 2001 Feb 13;98(4):2089-94. doi: 10.1073/pnas.98.4.2089. Epub 2001 Feb 6. PMID 11172080
- [Derived] Ure A, Cox GR, Haslam R, Williams K. Acetylcholinesterase inhibitors for autistic spectrum disorders. Cochrane Database Syst Rev. 2023 Jun 1;6(6):CD013851. doi: 10.1002/14651858.CD013851.pub2. PMID 37267443